CLINICAL TRIAL: NCT05666427
Title: Investigation of the Effect of Pelvic Floor Muscle Training Combined With Stabilization Exercises on Pain and Urinary Parameters in Individuals With Low Back Pain With Urinary Incontinence
Brief Title: Investigation of the Effects of Stabilization Exercises and Pelvic Floor Muscle Training on Pain and Urinary Parameters in Individuals With Chronic Low Back Pain With Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Ibrahim Kucukcan, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Kalyoncu-kucukcan001
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain; Urinary Incontinence
Keywords: low back pain; Urinary Incontinence; pelvic floor muscle training; stabilization exercises
MeSH Terms: conditions — Low Back Pain; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No application will be made until the end of this group work. After the end of the study, the effective protocol will be applied.
- Classic Application Group (Active Comparator): In this group, classical pelvic floor muscle training will be applied.
  Interventions: Behavioral: Pelvic floor muscle training
- Study Group (Active Comparator): The protocol determined for the study will be applied in this group. This protocol is planned as follows: It will perform stabilization exercises with the activation of the pelvic floor muscles.
  Interventions: Behavioral: Pelvic floor muscle training combined with stabilization exercises

INTERVENTIONS:
Behavioral: Pelvic floor muscle training combined with stabilization exercises — While people are doing stabilization exercises, they will also work the pelvic floor muscles. Practices will be combined with breathing.
  Arms: Study Group
Behavioral: Pelvic floor muscle training — Exercises that activate the pelvic floor muscles to strengthen and increase endurance.
  Arms: Classic Application Group

SUMMARY:
The research will be done with people with urinary incontinence and low back pain. 3 groups of volunteer participants will be formed. The groups were planned as study group, classical application group and control group. Classical pelvic floor muscle training will be applied to the classical application group. Pelvic floor muscle training combined with stabilization exercises will be applied to the study group. In this study, the effect of pelvic floor muscle training combined with stabilization exercises on pain and urinary parameters compared to classical pelvic floor muscle training will be investigated in people with urinary incontinence and low back pain at the same time.

DETAILED DESCRIPTION:
The rehabilitation period in the study was determined as 2 months. Participants will receive treatment with a supervisor 1 or 2 days a week. On other days, they will continue as a home program.

ELIGIBILITY:
Inclusion Criteria:

* Those with low back pain for at least 3 months (at least once a week with low back pain)
* Those with urinary incontinence
* 4 and above according to Numerical Pains Rating Scale
* At least 20% according to the Oswestry Disability Index
* Body Mass Index 30 and below

Exclusion Criteria:

* Those who have undergone lumbar or pelvic surgery in the last 6 months
* Those who received pelvic floor muscle training in the last 3 months
* Systemic, inflammatory, rheumatic, malignant, osseous pathologies etc. that may cause low back pain. those with diseases
* Those who are pregnant
* Stage 3-4 of pelvic organ prolapse
* Those who are pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | a day before rehabilitation
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'
Euro Quality of Life 5D-3L | a day before rehabilitation
  The EQ-5D-3L (European Quality of Life 5 Dimensions 3 Level Version) is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease
Incontinence Severity Index | a day before rehabilitation
  The incontinence severity index (ISI) consists of two questions, regarding frequency and amount of leakage. It categorizes urinary incontinence (UI) into slight, moderate, severe, and very severe.

SECONDARY OUTCOMES:
Modified Oxford Scale | a day before rehabilitation
  The Modified Oxford Scale (MOS) was used to rate pelvic floor muscle contraction on a scale of 0-511: 0 = no contraction; 1 = minor muscle 'flicker'; 2 = weak muscle contraction; 3 = moderate muscle contraction; 4 = good muscle contraction and 5 = strong muscle contraction
Tampa Kinesiophobia Scale | a day before rehabilitation
  The Tampa Scale of Kinesiophobia (TSK) that was developed in 1990 is a 17 item scale originally developed to measure the fear of movement related to chronic lower back pain.
Oswestry Disability Index | a day before rehabilitation
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.
Pain Catastrophizing Scale | a day before rehabilitation
  Pain catastrophizing is characterized by the tendency to magnify the threat value of a pain stimulus and to feel helpless in the presence of pain, as well as by a relative inability to prevent or inhibit pain-related thoughts in anticipation of, during, or following a painful event.
State-Trait Anxiety Inventory | a day before rehabilitation
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Higher scores are positively correlated with higher levels of anxiety. Its most current revision is Form Y and it is offered in more than 40 languages
Incontinence Quality of Life Instrument | a day before rehabilitation
  The I-QOL has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarrassment (5 items). It is easily self-administered and takes about 5 minutes to complete.
Urinary Distress Inventory | a day before rehabilitation
  The Urogenital Distress Inventory (UDI-6) is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Yakut, Professor, Study Director — Hasan Kalyoncu University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322